CLINICAL TRIAL: NCT05232136
Title: Oncolytic Virus (OH2) Adjuvant Therapy After Transurethral Resection of Bladder Tumor in Non-Muscle-Invasive Bladder Cancer Who Have Failed First-line Prophylactic Intravesical Instillation Therapy: a Phase Ⅰb/Ⅱ Clinical Trial
Brief Title: OH2 Oncolytic Viral Therapy in Non-Muscle-Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-016
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: Oncolytic Virus
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OH2 (Experimental): This arm include two doses (1x10e6, 1x10e7 CCID50/mL) of OH2 injection，the 1x10e6 CCID50/mL dose group should be delivered before the 1x10e7 CCID50/mL dose group.
  Interventions: Biological: OH2 injection

INTERVENTIONS:
Biological: OH2 injection — OH2: Oncolytic Type 2 Herpes Simplex Virus

SUMMARY:
This phase Ⅰb/Ⅱ study evaluates the safety and efficacy of OH2 for adjuvant therapy in non-muscle-invasive bladder cancer after first-line prophylactic intravesical instillation therapy.

OH2 is an oncolytic virus developed upon genetic modifications of the herpes simplex virus type 2 strain HG52, allowing the virus to selectively replicate in tumors. Meanwhile, the delivery of the gene encoding human granulocyte macrophage colony-stimulating factor (GM-CSF) may induce a more potent antitumor immune response.

DETAILED DESCRIPTION:
This is a phase Ⅰb/Ⅱ study evaluating the safety and efficacy of OH2 in non-muscle-invasive bladder cancer.

BH-OH2-016 is a single-arm,multicenter clinical trial. After screening, The treatment period includes induction treatment period and maintenance treatment period. In the induction treatment period, OH2 will be delivered once two weeks. In the maintenance treatment period, OH2 will be delivered once a month. In this trial, two doses (1x10e6, 1x10e7 CCID50/mL) of OH2 will be delivered intravesical instillation，and the 1x10e6 CCID50/mL dose group should be delivered before the 1x10e7 CCID50/mL dose group.

Adverse events (AEs) are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).Urine cytology/Cystoscopy/ultrasonography of urinary system will be used for disease recurrence examination.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 80 years old (including boundary value), male or female.
2. Failed in first-line preventive bladder perfusion therapy, and retained the bladder (or other reasons are not suitable for radical total cystectomy).
3. Ta, T1 or Tis with high grade (HG) of non-muscle-invasive bladder cancer.
4. Negative histology and pathology of bladder mucosa biopsy and negative postoperative urine cytology during TURBT.
5. No tumor was found in upper urinary tract examination; No systemic chemotherapy or radiation therapy for bladder cancer has been done at any time before.
6. ECOG 0-1.
7. The estimated survival time is more than 1 year.
8. Laboratory inspection:

   1. WBC≥3.5 × 10^9／L，ANC≥1.5 × 10^9／L，PLT≥80 × 10^9／L，Hb≥90g/L；
   2. Blood bun and serum creatinine were within 1.5 times of the upper limit of normal value;
   3. TBIL ≤ 1.5 times the upper limit of normal value;
   4. ALT and AST ≤ 2.5 times the upper limit of normal value;
   5. The coagulation function is normal (PT and APTT are within 1.5 times of the upper limit of normal value).
9. Received effective contraception during and within 3 months after treatment.
10. At least 3 months after the end of herpes infection.
11. Voluntary signing of informed consent, expected patient compliance

Exclusion Criteria:

1. muscle invasive bladder cancer or bladder cancer with clinical metastasis.
2. Complications occurred after TURBT, or perfusion therapy could not be performed.
3. Allergic to GM-CSF products or have a history of allergic reaction to the main and auxiliary materials of any dosage form in the study drug.
4. Suffering from serious medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, severe infection, active gastrointestinal ulcer.
5. Chemotherapy or radiotherapy is expected to be used during the study.
6. Active infection or fever of unknown cause > 38.5 ℃ during screening and before the first administration. Ongoing urinary system infection, especially bladder infection (if the infection can be controlled by antibiotics, except that it can return to normal after 7 days of antibiotic withdrawal).
7. Congenital or acquired immune deficiency (such as HIV infection) , Hepatitis B infection of HBV-DNA or more than 10 /mL, HCV antibody and HCV RNA positive in hepatitis C infection.
8. Pregnant or lactating.
9. Other experimental drugs or antiviral therapy were used or are being used within 4 weeks before treatment.
10. Participated in immunosuppressive therapy in recent 3 months, including cyclosporine, antithymocyte globulin or tacrolimus.
11. Participated in cancer vaccine treatment trials in recent 12 months (such as dendritic cell therapy and heat shock vaccine).
12. History of psychotropic substance abuse, alcoholism or drug abuse.
13. Other malignant tumors within 5 years before enrollment, except effectively resected cervical carcinoma in situ, low-risk gastrointestinal stromal tumor, skin basal cell carcinoma, skin squamous cell carcinoma, thyroid papillary carcinoma and breast ductal carcinoma in situ.
14. Active autoimmune diseases or history of autoimmune diseases and may relapse, except:

    1. Type I diabetes mellitus;
    2. Hypothyroidism (if only controlled by hormone replacement therapy);
    3. Controlled celiac disease;
    4. Skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, hair loss);
    5. Any other disease that will not recur without external triggers.
15. Using corticosteroids within 14 days before the administration of the study drug due to treatment, or suffering from any disease requiring systemic treatment with other immunosuppressants, except:

    1. Local, ophthalmic, intra-articular, intranasal or inhaled corticosteroids with minimal systemic absorption;
    2. Prophylactic short-term use of corticosteroids (e.g., allergy to contrast agents) or for the treatment of non autoimmune diseases (e.g., delayed hypersensitivity caused by contact allergens).
16. Not suitable to participate study judged by investigators for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
AEs | 1 years
  All events with a Grade 3 or above toxicity (defined by the CTCAE v5.0) will be tabulated by event and by relationship to OH2.
Relapse Free Survival Rate at 6 months | 6 months
  The assessment result is the number and proportion of subjects with relapse free survival at 6 months.
Relapse Free Survival Rate at 12 months | 12 months
  The assessment result is the number and proportion of subjects with relapse free survival at 12 months.
Rate of disease progression | 1 years
  Time after OH2 administration to clinical and radiographic disease progression will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China